CLINICAL TRIAL: NCT03238885
Title: Predicting Pathological Complete Response of Rectal Cancer to Neoadjuvant Chemoradiotherapy With MR Radiomics Method
Brief Title: Predicting Pathological Complete Response of Rectal Cancer With Magnetic Resonance(MR) Radiomics
Status: Completed | Type: Observational
Sponsor: Sun Ying-Shi (Other)
Responsible Party: Sponsor-Investigator, Sun Ying-Shi, Director, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Other Study IDs: RCpCR-MR-Radiomics
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LARC-CRT: LARC patients who will receive neoadjuvant CRT before surgical resection.
  Interventions: Diagnostic Test: pelvic MR examination

INTERVENTIONS:
Diagnostic Test: pelvic MR examination — All patients will take pelvic MR examination within 1 week before CRT and within 1 week before surgery.Pre- and post-CRT MRI examinations will be performed using a 3.0 T unit (Discovery 750) using an 8-channel phased array body coil in the supine position. To reduce colonic motility, 20mg of scopolamine butylbromide will be injected intramuscularly 30 min before MRI.

SUMMARY:
This study plans to construct a MR radiomics model for predicting pathological complete response(pCR) to neoadjuvant chemoradiotherapy(CRT) in locally advanced rectal cancer(LARC) patients.

DETAILED DESCRIPTION:
We propose to develop and validate a radiomics model for individualized pCR evaluation after CRT in patients with LARC. We plan to use both pre- and post-CRT MRI data to construct the predictive radiomics model for evaluating if LARC patients achieve pCR after CRT. The ultimate aim is to select appropriate LARC patients for omission of surgery.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proved rectal cancer
* locally advanced rectal cancer (≥T3 or N+)
* a distance less than 12cm between the lower edge of tumor and the anal margin
* no evidence of distant metastases
* no prior anti-cancer therapy before treatment
* scheduled to receive preoperative CRT

Exclusion Criteria:

* history or concurrent of other malignancy
* incomplete preoperative CRT
* failed to receive surgery or unavailable pCR assessment
* poor quality of MR images for measurement
* patient quit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: LARC patients who will undergo neoadiuvant CRT before surgery.
Sampling Method: Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Pathological complete response(pCR) | within one week after surgery
  Pathological complete response was defined as the absence of viable tumor cells in the primary tumor and lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Shi Sun, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No